CLINICAL TRIAL: NCT07080125
Title: Non-interventional Post-authorization Effectiveness Study to Assess Long-term Outcomes of Nintedanib Treatment in Patients With Systemic Sclerosis Associated Interstitial Lung Disease (SSc-ILD)
Brief Title: A Study Using a Disease Registry to Observe the Long-term Effects of Nintedanib in People With Scleroderma-related Lung Fibrosis
Status: Active, not recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0421; EUPAS106792 (Registry Identifier: EMA RWD catalogue)
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Interstitial Lung Diseases; Systemic Sclerosis Associated Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Individuals that initiate Ofev® including either:
  1. with an ongoing or new immunosuppressive therapy (IST) regimen (i.e., Ofev® combination therapy) or
  2. after discontinuing an IST regimen or individuals that have never been on IST (i.e. Ofev® monotherapy)
  Interventions: Drug: Ofev®
- Unexposed group: Individuals that do not initiate Ofev® during the study period and can include the following:
  1. Individuals on an IST regimen, described as 1a) those without an IST treatment escalation and 1b) those with an IST treatment escalation (i.e., increased dose, additional IST, switch in IST) to treat ILD- or non-ILD related SSc organ manifestations (e.g., mycophenolate, cyclophosphamide, methotrexate, tocilizumab, rituximab, etc.)
  2. Individuals who receive no IST

INTERVENTIONS:
Drug: Ofev® — Ofev®
  Other Names: Nintedanib
  Groups: Exposed group

SUMMARY:
This post-approval registry study is planned to generate data to address remaining questions on long-term effectiveness and to better characterize longer term beneficial effects of Nintedanib in patients with systemic sclerosis associated interstitial lung disease (SSc-ILD) in terms of survival, quality of life, pattern of disease progression as well as effectiveness and safety in the subgroup of patients with pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the EUSTAR registry
* Provided consent at their site to have their data included in the EUSTAR registry for a broad range of research studies, and agree to visit the site every 12 months
* Have a diagnosis of ILD defined by radiological findings on High Resolution Computed Tomography (HRCT) and/or X-ray that is documented in the electronic Case Report Form (eCRF) by the treating physician

Exclusion Criteria:

* Women with Systemic Sclerosis Interstitial Lung Disease (SSc-ILD) who are pregnant, or breastfeeding will be excluded since Ofev® is contraindicated for women who are pregnant due to safety concerns
* SSc-ILD patients aged <18 years: only adults will be included in the study since Ofev® is approved for treatment of SSc-ILD in adults
* Patients with a previous Hematopoietic Stem Cell Transplantation (HSCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will constitute patients with Systemic Sclerosis (SSc) and Interstitial Lung Disease (ILD) (based on radiological evidence) enrolled in the European Scleroderma Trials and Research (EUSTAR) registry.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to absolute Forced Vital Capacity (FVC) decline (% predicted) ≥5%, lung transplantation (indicating end stage ILD), or death | up to 10 years
Time to absolute FVC decline (% predicted) ≥10%, lung transplantation (indicating end-stage ILD), or deat | up to 10 years

SECONDARY OUTCOMES:
Time to absolute (% predicted) FVC decline ≥5% | up to 10 years
Time to absolute (% predicted) FVC decline ≥10% | up to 10 years
Time to relative (ml) FVC decline ≥5% | up to 10 years
Time to relative (ml) FVC decline ≥10% | up to 10 years
Time to lung transplantation (indicating end-stage ILD) | up to 10 years
Time to death | up to 10 years
Change from baseline in FVC (% predicted) | at baseline, up to 10 years
Change from baseline in FVC (ml) | at baseline, up to 10 years
Lung specific Quality of Life (QoL) measured as change from baseline of total, impact, and symptom scores using the Living with Pulmonary Fibrosis (L-PF) questionnaire, measured as change of baseline at years 1, 2, 3,….10 | at baseline, up to 10 years
  The L-PF patient reported outcome measure (PROM) is a questionnaire designed for patients with fibrosing ILDs and developed with those patients to investigate their level of symptoms and QoL.
  The L-PF consists of two modules, symptoms and impacts, and five scales: symptoms total, dyspnea, cough, fatigue, impacts total, and Total L-PF score.
  Items in both modules have response options on a five-option numeric rating score with an anchor of 0 "Not at all" to 4 "Extremely". Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.
Time to worsening of Pulmonary Hypertension (PH) in the sub-population of patients with PH at baseline | up to 10 years
  Worsening of PH is defined as a composite outcome of the following:
  1. time to all-cause death;
  2. time to non-planned PH-related hospitalization; or 3) time to PH-related deterioration identified by at least one of the following parameters: i. increase in World Health organization functional class, ii. deterioration in exercise testing; or iii. Signs or symptoms of right-sided heart failure
Incidence rate of major bleeding (defined as those requiring intervention or hospitalization) in exposed vs unexposed treatment groups | up to 10 years
Final outcome for the major bleeding events (i.e., recovered or fatal) overall | up to 10 years
Proportion of patients with major bleeding that had a pre-existing risk for bleeding | up to 10 years
Incidence rate of gastrointestinal perforations in exposed vs unexposed treatment groups | up to 10 years
Final outcome (i.e., recovered or fatal) for gastrointestinal perforation events overall | up to 10 years
Proportion of patients with gastrointestinal perforations that had a pre-existing risk for gastrointestinal perforations | up to 10 years
Incidence rate of thromboembolism (arterial or venous) in exposed vs unexposed treatment groups | up to 10 years
Final outcome (i.e., recovered or fatal) for thromboembolic events overall | up to 10 years
Proportion of patients with thromboembolism that had a pre-existing risk for thromboembolism | up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- EUSTAR Registry, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com